CLINICAL TRIAL: NCT05329753
Title: Effectiveness of a Mobile Health Intervention for the Prevention of Overweight and Obesity in Adolescents on Sport and Nutrition Knowledge, Eating Habits and Physical Activity: A Randomized Clinical Trial
Brief Title: Effectiveness of a Mobile Health Intervention for the Prevention of Overweight and Obesity in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI-77.18 EIESOJTIC18
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Adolescent Obesity
Keywords: mobile application; eating habits; physical activity; overweight; nutrition knowledge
MeSH Terms: conditions — Pediatric Obesity; Feeding Behavior; Motor Activity; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Mobile application
  Interventions: Device: Mobile health application
- Control group (No Intervention): Usual education

INTERVENTIONS:
Device: Mobile health application — Health intervention through a smartphone application that favors the process of learning
  Arms: Intervention group

SUMMARY:
The prevention of overweight and obesity in adolescents is a public health priority given the impact of obesity on both short- and long-term health. Scientific evidence has shown that interventions in diet and physical exercise can reduce the risk of obesity in children and young people since adolescence is an ideal stage for educating on a healthy lifestyle and correcting the habits that may have been acquired in childhood. Smartphone applications (apps) can provide a useful alternative to overweight and obesity prevention measures.

The objective of this study was to evaluate, through a randomized controlled clinical trial, the effect of an intervention based on a mobile health application (m-Health) on improving the degree of sport and nutrition knowledge, eating habits, and level of physical activity of adolescents.

The sample consists of 305 adolescents, 154 in the intervention group and 151 in the control group that are evaluated at the beginning and 6 months later regarding sociodemographic, eating habits, food knowledge, level of physical activity, body mass index, and waist circumference. The educational intervention was carried out using an m-Health tool, a mobile phone application. The outcomes were changes in the mentioned variables to a six-month follow-up between the two groups.

DETAILED DESCRIPTION:
Design: A randomized parallel-group, controlled clinical trial was performed on adolescents from public secondary schools in the province of Cadiz, Spain.

Randomization and Blinding: The randomization and allocation to each group (1:1, intervention, and usual care) are based on computer-generated random numbers stratified in the three courses of secondary education. The researchers responsible for the study do not participate in the allocation of the participants. Due to the kind of intervention, blinding is not possible when the participants are allocated to groups. To minimize any bias, objective clinical variables are measured during the evaluation visit and the analyses are performed by blinded researchers.

Study Sample: The estimated sample size to detect a mean difference of at least one point in the level of healthy eating habits, measured by the KidMed questionnaire, with a standard deviation of the values in the questionnaire known from previous studies of 2.5 points, a level of confidence of 95% and statistical power of 90%, it was 126 participants in each group, intervention, and control. Assuming a 20% loss to follow-up, 305 participants were recruited, 154 in the intervention group and 151 in the control group.

Recruitment: All participants, in the intervention and control groups, received an Intervention on healthy habits consisting of four sessions developed by a nurse over two months. Adolescents who voluntarily decided to participate in the mobile Health educational intervention were recruited by a nurse. Both the adolescents and their parents signed the informed consent.

Intervention: The nurse installs the application on the mobile phone of the participants in the intervention group. It is a friendly, easy-to-use application for smartphones and tablets that favors the process of learning while playing.

Application Contents: Through the application, the adolescent participates in five activities: food, exercises, tests, learning more, and games that are different from each other but interconnected and that allow progress to be seen. The application "Care your habits" has educational materials on nutrition and physical activity. The participant records the food eaten and the physical activity performed, in addition to answering health questionnaires.

Technical Data of the Application:

The application has been developed for Android mobiles with versions between API 16 and API 28, which guarantees user compatibility. This app uses Firebase, a cloud platform that enables certain features, such as a secure login for app users. The application uses an initial Activity, which is responsible for managing the Login. The application is structured in different Fragments. Each of these Fragments is made up of a layout that is the graphical interface that the user sees and a class in the Java programming language that is the part in charge of processing the user's interaction with the interface and performing the appropriate action.

The app needs a server that manages interactions with the database where the data that users provide voluntarily from the app itself is stored. The part of the server that supports and complements the Android application is made up of a RESTful API developed in the NodeJS programming language. This server communicates with Firebase in order to verify the identity of the user who is providing data at all times, so that a user could not falsify another user's data.

All of this information is persistently stored in a NoSQL database, specifically a MongoDB database. The information provided by users is encrypted to prevent data theft.

Ethical Considerations: The study was conducted in agreement with the guidelines and protocols established in the Helsinki Declaration as revised in Fortaleza (Brazil) in October 2013, and complies with Law 14/2007 on Biomedical Research and with European Data Protection Regulations. The Biomedical Research Ethics Committee of Cádiz, Andalusian, approved the project with the reference: 11_02_2019. The informed written consent of all the participants and their parents was requested. The application guarantees security measures regarding the current General Data Protection Regulations in Europe. It also includes data encryption mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents who were studying the 1st to 3rd grades of secondary education in public institutes
* Have a smartphone or tablet with an Android operating system and internet access

Exclusion Criteria:

* Adolescents with barriers that prevented them from understanding the characteristics of the study: Comprehension, visual or auditory problems
* Adolescents with disease or treatment that affect the variables studied (diagnosed diseases that affect body weight such as liver or kidney disease or regular treatment with drugs such as corticosteroids)

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 305 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Eating habits | 6 months
  KidMed: A 16-item Questionnaire of Mediterranean diet adherence (unit of measure: points. Each item is scored 0 or 1. The total Mediterranean diet score ranges from 0 to 12 points. The higher the score, the higher the degree of adherence to the Mediterranean Diet).
Nutrition knowledge | 6 months
  General and Sport Nutrition knowledge Questionnaire: A questionnaire with 62 items (unit of measure: points. The higher the score, the higher the knowledge level)
Level of physical activity | 6 months
  Physical Activity Questionnaire for adolescents (PAQ-A) (The overall result of the test is a score from 1 to 5 points that allows to establish a graduation in the level of physical activity made by each adolescent. Do higher values represent a better outcome)

SECONDARY OUTCOMES:
Body mass index | 6 months
  Body mass index is calculated as weight in kilograms divided by height in meters squared. The WHO tables for adolescents by age and sex were used to classify the body mass index of adolescents as normal, overweight, and obese.
Waist circumference | 6 months
  Waist circumference was defined as the smallest abdominal circumference between the lowest rib and the upper anterior iliac spine.
  Percentile tables for Spanish adolescents by age and sex were used

CONTACTS AND LOCATIONS:
Overall Officials: M J Santi, MD, Principal Investigator — University of Cádiz
Locations (1):
- University of Cádiz, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No